CLINICAL TRIAL: NCT07086014
Title: Cue Reactivity Modulation in MSM With Methamphetamine Use Disorder
Brief Title: Methamphetamine Cue-reactivity
Status: Recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Muhammad Parvaz, Associate Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: STUDY-20-00284; R61DA056779 (NIH)
Record Dates: First submitted 2025-07-18; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Methamphetamine Use Disorder
Keywords: methamphetamine; cue-reactivity; craving; EEG; incubation; cognitive reappraisal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- MSM - MUD (Current): Participants who are MSM and are currently using methamphetamine (MA abstinence: 2 weeks; range: 1-3 weeks).
  Interventions: Behavioral: Cognitive Reappraisal
- MSM - MUD (Abstinent): Participants who are MSM and are abstaining from using methamphetamine (MA abstinence: 3 months; range: 2-4 months).
  Interventions: Behavioral: Cognitive Reappraisal
- non-MSM - MUD (Current): Participants who are not MSM and are currently using methamphetamine (MA abstinence: 2 weeks; range: 1-3 weeks).
  Interventions: Behavioral: Cognitive Reappraisal
- non-MSM - SUD (Abstinent): Participants who are not MSM and are abstaining from using methamphetamine (MA abstinence: 3 months; range: 2-4 months).
  Interventions: Behavioral: Cognitive Reappraisal

INTERVENTIONS:
Behavioral: Cognitive Reappraisal — an emotion-regulation strategy while being asked to complete cognitive tasks.

SUMMARY:
In this observational cohort study, the researchers propose to first identify a psychophysiological marker of methamphetamine cue-reactivity and its incubation with abstinence from methamphetamine use (MUD) and examine group-differences between men who have sex with men (MSM) and non-MSM MUD.

The primary objective is to identify psychophysiological markers of methamphetamine (MA) cue-reactivity and its abstinence incubation. The secondary objective is to examine group-differences in methamphetamine use disorder (MUD) individuals between homosexual men (MSM) and heterosexual men (non-MSM). The primary endpoint is to assess incubation of cue-reactivity longitudinally with its reduction in cognitive reappraisal, and the secondary endpoint is to examine the impact of cognitive reappraisal on clinical outcomes of methamphetamine use disorder (MUD) in homosexual men (MSM).

2-year long study. Screening and enrollment will be done at different locations of the Addiction Institute of Mount Sinai. The EEG session will be done at Icahn School of Medicine at Mount Sinai. Participation in the research study will be for a single EEG session.

DETAILED DESCRIPTION:
Cognitive Reappraisal (CR) is an extensively characterized emotion-regulation strategy that impacts early cognitive stages of emotion-generative processes and can be used to regulate emotional experience and expression. CR techniques include "distancing" that aims at changing the emotional impact of a situation by taking the perspective of a detached observer, and "reinterpretation" that focuses on re-evaluating the emotional situation in unemotional terms. Neuroimaging studies of CR implicate the engagement of regions that have typically been associated with conflict monitoring, selective attention, and regulation of negative affect. A growing literature indicates that CR can attenuate heightened cue-reactivity in addicted individuals. The researchers preliminary data in CUD are consonant with this view and show that decrease in cue-reactivity can be quantified by a reduction in the LPP (Parvaz et al., PNAS, 2021). The researchers have also shown that more frequent use of CR is correlated with reduced cue-reactivity and lower craving in CUD. Others have reported that CR can modulate attention bias to affective stimuli with sustained decrease even after regulation demands are lifted. Clinical studies show that CR training is associated with better cognitive control, and better clinical outcomes in smokers. Thus, CR has the potential to decrease MA cue-reactivity and may lead to better clinical outcomes in MSM with MUD.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and give informed consent
* Identify as either MSM or non-MSM
* Males; Age 18-60
* DSM-5 Diagnosis of MUD (Methamphetamine Use Disorder)
* Have appropriate abstinence duration [i.e., current Methamphetamine users (MA): 2 weeks (range: 1-3 weeks); MA-abstinent: 3 months (range: 2-4 months)]
* Treatment-seeking MUD must be in a treatment facility for substance use disorder, with MA as the primary drug (at the first visit)
* Treatment-seeking MUD must be abstinent from MA use for approximately 2 weeks (range: 1-3 weeks) at enrollment.

Exclusion Criteria:

• Women

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This is a study on MSM and non-MSM males only, who have shown to be at a high risk for methamphetamine use disorder.
Study Population: 44 current MA-using (MA abstinence: 2 weeks; range: 1-3 weeks), and 44 MA-abstinent (MA abstinence: 3 months; range: 2-4 months), individuals with MUD. Importantly, 50% in each group will be MSM, and the other 50% will be non-MSM men, resulting in 4 groups: (1) MSM/current MA, (2) MSM/abstinent, (3) non-MSM/current MA, and (4) non-MSM/abstinent; n=22 per group, matched on age and HIV status. Men who identify as "homosexual/gay" or "bisexual" and/or report having had sex with a man in the last 12 months will be defined as "MSM" and those who identify as "heterosexual/straight" and do not report having sex with men in the last 12 months as "non-MSM".
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in EEG-derived late positive potential (LPP) Amplitude | at approx. 2 weeks and 3 months abstinence
  Change in amplitude (or incubation of) the EEG-derived late positive potential (LPP) - an objective neurophysiological marker of drug cue-reactivity - occurs 400 msec after the onset of a drug-related cue. The LPP amplitude has also shown to predict self-reported craving, simulated drug-seeking behavior and relapse, highlighting the clinical utility of this objective metric of cue-reactivity.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad A Parvaz, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. Any purpose. Data are available indefinitely at (Link to be included in the URL field below).
URL: https://openneuro.org/